CLINICAL TRIAL: NCT06003309
Title: Frequency and E-field Enhancement of ITBS for Depression (FREED)
Acronym: FREED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Zafiris Daskalakis, Chair of Psychiatry Department, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 807836
Record Dates: First submitted 2023-07-11; First posted 2023-08-21 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- The fully individualized form of iTBS (BOTH the frequency and E-field targeting approaches) (Active Comparator): In the Ind-iTBS, the coil placement and current amplitude will be provided using individualized E-field modeling and coordinate-based cortical targeting. The stimulation frequency will also be individualized according to EEG-derived TGC.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) - Fully Individualized iTBS
- iTBS individualized using E-field targeting only (targeted-iTBS) (Active Comparator): In the targeted-iTBS, the coil placement and current amplitude will be provided using individualized E-field modeling and coordinate-based cortical targeting.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) - targeted-iTBS
- Standard iTBS treatment (i.e., typical iTBS localized to the DLPFC using the Beam F3 method) (Active Comparator): The standard iTBS will be delivered with the typical 5Hz/50Hz patterned frequencies used in the FDA-approved treatment protocol and stimulation will be delivered according to the Beam F3 targeting.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) - Standard-iTBS

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) - Fully Individualized iTBS — Repetitive transcranial magnetic stimulation (rTMS) is a safe and effective treatment for TRD that is increasingly being used in clinical practice across the world. It's mechanism of action is based on Farady Law of electromagnetic induction where the magnetic field produced by TMS coil induces electric field in the neurons. In the Ind-iTBS, the coil placement and current amplitude will be provided using individualized E-field modelling and coordinate-based cortical targeting. The stimulation frequency will also be individualized according to EEG-derived TGC.
  Arms: The fully individualized form of iTBS (BOTH the frequency and E-field targeting approaches)
Device: Transcranial Magnetic Stimulation (TMS) - targeted-iTBS — Repetitive transcranial magnetic stimulation (rTMS) is a safe and effective treatment for TRD that is increasingly being used in clinical practice across the world. It's mechanism of action is based on Farady Law of electromagnetic induction where the magnetic field produced by TMS coil induces electric field in the neurons. In the targeted-iTBS, the coil placement and current amplitude will be provided using individualized E-field modelling and coordinate-based cortical targeting.
  Arms: iTBS individualized using E-field targeting only (targeted-iTBS)
Device: Transcranial Magnetic Stimulation (TMS) - Standard-iTBS — Repetitive transcranial magnetic stimulation (rTMS) is a safe and effective treatment for TRD that is increasingly being used in clinical practice across the world. It's mechanism of action is based on Farady Law of electromagnetic induction where the magnetic field produced by TMS coil induces electric field in the neurons. The standard iTBS will be delivered with the typical 5Hz/50Hz patterned frequencies used in the FDA approved treatment protocol and stimulation will be delivered according to the Beam F3 targeting.
  Arms: Standard iTBS treatment (i.e., typical iTBS localized to the DLPFC using the Beam F3 method)

SUMMARY:
The investigators propose a randomized 3-arm double-blinded parallel experimental trial (20 sessions over 4 weeks) in 75 patients with TRD. The three arms include (1) the combination of a fully Individualized form of intermittent Theta Burst Stimulation (iTBS) (using BOTH the frequency and electric field (E-field) targeting approaches) (Ind-iTBS)), (2) iTBS individualized using E-field targeting only (targeted-iTBS) and (3) Standard iTBS treatment (i.e., typical iTBS localized to the dorsolateral prefrontal cortex (DLPFC) using the Beam F3 method). Electroencephalography (EEG) data will be collected at rest and during a working memory task, at baseline, and at the end of treatment along with clinical assessments of depression severity. The target engagement dependent variable of interest in these three arms will be fronto-parietal theta connectivity measured through resting-state EEG. The investigators hypothesize that stimulation with Ind-iTBS will lead to greater changes in fronto-parietal theta connectivity than that produced with targeted-TBS and standard iTBS. Aim: To evaluate the effects of two individualized forms of iTBS (i.e., using BOTH the frequency and E-field individualization; Ind-iTBS) compared to iTBS individualized for E-field targeting only (targeted-iTBS) and standard iTBS on fronto-parietal theta connectivity. Hypotheses: (1) Ind-iTBS will lead to greater changes in fronto-parietal theta connectivity compared to both targeted-iTBS and standard iTBS. (2) Ind-iTBS will also lead to a greater reduction in depressive symptoms (as defined by the mean reduction in Montgomery Åsberg Depression Rating Scale Scores (MADRS)) compared to both targeted-iTBS and standard iTBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive episode (MDE, in accordance with the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5), in the context of unipolar major depressive disorder disorder.
* 18-80 years of age.
* Male or female.
* At least one failed antidepressant medication trial at level 3 in the Antidepressant Treatment History Form: Short Form (ATHF-SF) classification.
* Montgomery-Asberg Depression Rating Scale (MADRS) Score of >19 (moderate - severe depression).
* No increase or initiation of new antidepressant therapy in the four weeks prior to screening.
* Demonstrated capacity to give informed consent.

Exclusion Criteria:

* Inability to provide informed consent.
* Medically unstable patients.
* Concomitant neurological disorder or a history of a seizure disorder.
* Patients who are pregnant or breastfeeding.
* Any psychotic disorder or current active psychotic symptoms.
* Patients who have intracranial implants, other medical device or condition deemed unsafe for TMS.
* Contraindication to MRI scanning.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from pre-treatment in fronto-parietal theta connectivity at post-treatment | pre-treatment (within 24 hours prior to first treatment) and post-treatment (within 72 hours of final treatment)
  Source-localized fronto-parietal theta connectivity will be calculated from resting EEG

CONTACTS AND LOCATIONS:
Locations (2):
- University of California, San Diego, La Jolla, California, United States
- Australian National University, Canberra, Australia

IPD SHARING:
Plan to Share IPD: No